CLINICAL TRIAL: NCT03363490
Title: The Study of Neuromuscular Exercise Therapy and Patients Self-management Program in Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Jishuitan Hospital (Other); General Hospital of Beijing PLA Military Region (Other); Peking Union Medical College Hospital (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Lin Jianhao, Clinical Research Center of Osteoarthritis, Peking University People's Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PLSKNLSMFS2
Record Dates: First submitted 2017-11-26; First posted 2017-12-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Exercise Therapy
Keywords: Self-Management; Neuromuscular Exercise Therapy; Knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Self-Management

STUDY DESIGN:
Intervention Model Description: Patients of knee OA will be divided into A, B, C, D four parallel groups with fully informed, each group will enroll 100 patients, A for control group, B for neuromuscular exercise, C for self-management program, D for neuromuscular exercise and self-management program, respectively.
Who Masked: Outcomes Assessor
Masking Description: Assessor will not know which group the patients are enrolled when evaluate the baseline and follow-up situation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Other): The patients in this group will only receive health education intervention.
  Interventions: Behavioral: Health education
- Neuromuscular exercise therapy (Other): The patients in this group will receive exercise therapy intervention.Besides, health education will be performed for every group.
  Interventions: Behavioral: Neuromuscular exercise therapy; Behavioral: Health education
- Self-management program (Other): The patients in this group will receive self-management intervention.Besides, health education will be performed for every group.
  Interventions: Behavioral: Self-management program; Behavioral: Health education
- Exercise therapy+self-management (Other): The patients in this group will receive exercise therapy and self-management intervention.Besides, health education will be performed for every group.
  Interventions: Behavioral: Self-management program; Behavioral: Neuromuscular exercise therapy; Behavioral: Health education

INTERVENTIONS:
Behavioral: Self-management program — Self-management diary will record the frequency of pain, fatigue and injury of knee joint due to knee OA, if patients maintain proper activities, it will be also recorded by an smart phone APP. Patients diet and intake calorie will also be recorded in the diary，which help clinicians to adjust their diet, control their body weight.
  Arms: Exercise therapy+self-management; Self-management program
Behavioral: Neuromuscular exercise therapy — The exercise therapy is basically combined with neuromuscular training and anti resistance training. The aim is to improve the stability of the joints, enhance sensory motor control of lower extremities, reconstruct neutral position line. The exercise mode, frequency, intensity and duration will be adjusted individually through monitoring patient's pain.
  Arms: Exercise therapy+self-management; Neuromuscular exercise therapy
Behavioral: Health education — All four groups of patient will receive two times of health education in the first week.

SUMMARY:
Osteoarthritis is the most common chronic disabling disease,the importance of patient's self-management in chronic disease has been paid more and more attention internationally. Currently, the self-management of OA patients in China is lack of instructions from professional clinicians, and leads to inappropriate excise, irregular drug medication. OAKP (Osteoarthritis of the Knee Self-Management Program) is a program initiated from University of Southern Denmark, follows clinical guidelines of OA, formatted for easy use by patients and clinicians, including customized neuromuscular exercise therapy, educational sessions of what is OA and how to control body weight to protect the knee.

The main purpose of this study is to verify the effectiveness of neuromuscular exercise therapy and OAKP, see whether it can help patients to relief the symptom and improve life quality.

DETAILED DESCRIPTION:
The study plans to enroll patients above 50 years old who suffered from knee OA, but patients meets any of the exclusion criteria will not be enrolled. 400 patients of knee OA will be randomly divided into A, B, C, D four parallel groups with fully informed, each group will enroll 100 patients, A for control group, B for neuromuscular exercise, C for self-management program, D for neuromuscular exercise and self-management program, respectively. Each collaborate hospital would enroll patients as a multicenter clinical trial. Patient will receive a baseline and 3m, 6m, 12m follow-up evaluation of their knee physical function. Primary outcome measure is KOOS (Knee Injury and Osteoarthritis Outcome Score), secondary evaluation include VAS, EQ-5D, Arthritis self-efficacy score, 6-minutes Walk test, TUG test, 20 meters quick walk test,Stand up test in 30 seconds, Balance test, Kellgren& Lawrence（KL）, Pain medication. Outcome will compare the mean difference between baseline survey and 12 months of follow-up in each group, using t-test or chi-square test,respectively.

ELIGIBILITY:
Inclusion Criteria:

-

1.Clinical diagnosis of knee osteoarthritis, Diagnostic criteria is based on the Chinese medical association's 2007 diagnosis and treatment guidelines for osteoarthritis:

1. Repeated knee joint pain within 1 month;
2. X-ray(weight-bearing or not)shows narrowed joint space,sclerosis and (or) cystic degeneration of subchondral bone, osteophytes of the joints;
3. The joint fluid (at least twice) is clear and viscous, WBC<2000个/ml;
4. Age of patients ≥40 yrs;
5. Morning stiffness≤3 min;
6. Bone friction in the activity; Note：Combine clinical feature, laboratory and X-ray examination,when the patients meet(1)+(2) or (1)+(3)+(5)+(6) or (1)+(4)+(5)+(6)，they can be diagnosis as knee osteoarthritis.

2.VAS≥4分; 3.No surgical treatment is planned within 6 months;

Exclusion Criteria:

1. Other types of arthritis, such us RA(rheumatoid arthritis)
2. Severe deformity of knee joint;
3. Over obesity patients（BMI>35）;
4. Other comorbidities that would severely affect somatic function, such as: cerebral infarction, lumbar disease that meets surgical indications, lower extremity angiopathy;
5. Decompensated cardiac dysfunction;
6. Severe cardiovascular and cerebrovascular diseases, or the patient is too weak for any kinds of exercise;
7. Lack of compliance;

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
The Western Ontario and McMaster Universities Osteoarthritis Index，WOMAC | Baseline, 3 months, 6 months, 12months
  WOMAC grade is a reliable knee osteoarthritis patients' self-reported therapeutic effect evaluation system, including three dimensions: pain, stiffness, daily activities and quality of life, and each dimension includes several questions scale from 0(worst) to 4(best) , total score of each dimension range from zero (worst) to 100 (best). Score of each question add together will be the total score. Baseline, 3 months, 6 months, 12 months, through visit or telephone follow-up will be recorded. Compare the mean difference of WOMAC grade between baseline survey and 12 months of follow-up in each group.

SECONDARY OUTCOMES:
Visual Analog Score（VAS） | Baseline, 3 months, 6 months, 12months
  Visual Analogue Scale of pain is a scale to extimate pain, and its score ranges from 0(worst) to 10(best). The higher the score is, the more severe pain the patient is feeling.
EuroQol Five Dimensions Questionnaire（EQ-5D） | Baseline, 3 months, 6 months, 12months
  EQ-5D is a scale to extimate health condition and quality of life, and its score ranges from -0.6 to 1.0. The higher the score is, the healthier the patient is.
Kellgren& Lawrence（KL） | Baseline
  The higher the KL score is ,the more severe the patient is. Baseline,through visit or telephone follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhao Lin, MD, Principal Investigator — arthritic clinic and research center
Locations (1):
- PekingUPH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ageberg E, Roos EM. Neuromuscular exercise as treatment of degenerative knee disease. Exerc Sport Sci Rev. 2015 Jan;43(1):14-22. doi: 10.1249/JES.0000000000000030. PMID 25390299